CLINICAL TRIAL: NCT00588120
Title: Investigations Into the Genotype and Phenotype of Unclassified Hyperoxaluria: Enteric Oxalate Absorption Study
Brief Title: Enteric Oxalate Absorption Study in Unclassified Hyperoxaluria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Oxalosis and Hyperoxaluria Foundation (OHF) (Other)
Responsible Party: Principal Investigator, John Lieske, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1026-98; RFA-OD-08-001 (Other Grant/Funding Number: Rare Diseases Clinical Research Consortia); 1U54DK083908-01 (NIH)
Record Dates: First submitted 2007-12-26; First posted 2008-01-08 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Enteric Hyperoxaluria; Hyperoxaluria
Keywords: Hyperoxaluria; Unknown Hyperoxaluria; Enteric Hyperoxaluria; Oxaluric; High Oxalate; Oxalate; C13; Oxalate Diet
MeSH Terms: conditions — Hyperoxaluria | interventions — Oxalates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- C-13 labeled oxalate (Experimental): Hyperoxaluric patients
  Interventions: Drug: C-13 labeled oxalate

INTERVENTIONS:
Drug: C-13 labeled oxalate — A single prescribed dose of C-13 labeled oxalate will be given orally in capsule form or in jello. Urine will be collected for 24 hours after the dose.
  Take one capsule by mouth for one day.
  Other Names: oxalate

SUMMARY:
The purpose of this study is to learn more about a condition called 'unclassified hyperoxaluria'. People with this condition have large amounts of oxalate in their urine, which can cause kidney stones and kidney failure. We do not know what causes the high level of oxalate in the urine. In this study, we will evaluate absorption of a test dose of oxalate taken orally by measuring the amount of the test dose that is eliminated in the urine. We will compare the results of affected patients to healthy volunteers.

DETAILED DESCRIPTION:
Participants' oxalate intake and output will be monitored and assessed over a 24 hour period. Participants will ingest a prescribed oxalate dose and urine oxalate will be monitored for the 24 hour study period.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 4 years (patient must be able to void on request).
* Have good health.

Exclusion Criteria:

* Any prior history of renal disease, or hypertension
* ALL subjects (controls and affected patients) will be asked to discontinue any diuretics, calcium supplements, H2 blockers, proton pump inhibitors or gastrointestinal motility agents for approximately one week prior to initiation of the study.
* Subjects with GFR < 50 cc/min will be excluded.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 1998-12; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Urine oxalate measured following absorption of oral oxalate dose | 2 years
  Subjects with hyperoxaluria will be given an oral test dose of oxalate, with measurement of urine oxalate excretion over the next 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Milliner, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States